CLINICAL TRIAL: NCT03599206
Title: CXCL10/CXCR3 Regulation of Ozone-Induced Epithelial Permeability
Brief Title: ONES Grant: CXCL10/CXCR3 Regulation of Ozone-Induced Epithelial Permeability
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Robert Tighe, MD (Other)
Responsible Party: Sponsor-Investigator, Robert Tighe, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Pro00088966
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Environmental and Genetic Factors on Lung Function
Keywords: genetic: CXCR3 polymorphism rs2280964
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ozone (Experimental)
  Interventions: Drug: Ozone
- Filtered Air (Placebo Comparator)
  Interventions: Other: Filtered Air

INTERVENTIONS:
Drug: Ozone — Subjects will perform alternating 15 minutes rest with 15 minutes treadmill walk exercise periods for 135 minutes in while breathing Ozone (O3).
  Arms: Ozone
Other: Filtered Air — Subjects will perform alternating 15 minutes rest with 15 minutes treadmill walk exercise periods for 135 minutes in while breathing filtered air.
  Arms: Filtered Air

SUMMARY:
The purpose of this research study to understand how environmental and genetic factors may be involved in lung function. Study participants will undergo a 1-day screening that includes a blood draw and breathing testing, return for a two-day series of testing to include blood draw, and brief breathing test before and after an inhaled challenge with either filtered air (FA) or ozone (O3). Participants return the next day for a brief breathing test, a blood draw and a procedure called bronchoscopy to evaluate the lung after the challenge. Participants then return 18 - 20 days later to repeat the two-day series of testing to be challenged with the exposure not received on the first series, (FA or O3). Each visit will take about 3 - 3.5 hours. Follow-up phone calls from the study team will occur at 24 hours after each 2-day test series. Total study duration is about one to one-and a half months.

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment in the NIEHS Environmental Polymorphism Registry located in the greater Raleigh-Durham area
* Wild type or homozygous (female)/hemizygous (male - since sex-linked) expression of the CXCR3 polymorphism rs2280964

Exclusion Criteria:

* Current smokers of tobacco products including e-cigarettes or those with previous smoking history within the prior 5 years
* BMI less than 37 kg/m2
* Pregnant women and women who are presently lactating.
* Subjects that have received antibiotic administration or an upper respiratory infection within the previous 4 weeks
* College and graduate students or employees who are under direct supervision by any of the investigators in this protocol
* Alcohol or illicit substance abuse
* Chronic cardio/pulmonary respiratory disorders or other medical conditions as determined by the investigator
* Increased airway hyperresponsiveness at baseline as measured by a positive methacholine challenge response (methacholine PC20 FEV1 < 8 mg/ml)
* Subjects will be requested to refrain from antihistamines, nonsteroidal anti-inflammatory agents, antioxidants (e.g. beta-carotene, selenium, and lutein) and supplemental vitamins (e.g. C and E), for 1 week prior to, and during testing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Change in Ozone (O3) induced epithelial permeability, as measured by the level of clara cell secretory protein (ng/mL) | Baseline, 21 days
  This measure is defined by the comparing each individuals baseline (following filtered air challenge) to the ozone response. The investigators will perform two tests on this response as a means of confirmation. The individual will have blood drawn to obtain serum and a bronchoscopy to obtain bronchoalveolar lavage. The serum will be used to determine the level of clara cell secretory protein. This is measured by enzyme-linked immunosorbent assay (ELISA). The value is reported as ng/mL. Each value will be compared to the individuals filtered air control and reported as a fold change from baseline. These are independent values but are both accepted in the literature as measures of epithelial permeability.
Change in Ozone (O3) induced epithelial permeability, as measured by albumin level (ug/mL) | Baseline, 21 days
  This measure is defined by the comparing each individuals baseline (following filtered air challenge) to the ozone response. The investigators will perform two tests on this response as a means of confirmation. The individual will have blood drawn to obtain serum and a bronchoscopy to obtain bronchoalveolar lavage. The bronchoalveolar lavage will be similarly used to define the albumin level. Albumin is also measured by ELISA. The value is reported at ug/mL. Each value will be compared to the individuals filtered air control and reported as a fold change from baseline. These are independent values but are both accepted in the literature as measures of epithelial permeability.

SECONDARY OUTCOMES:
Change in Ozone O3 induced alterations in gene expression of airway epithelial cells, and bronchoalveolar lavage cells | Baseline, 21 days
  Measured by real-time PCR
Change in Ozone O3 induced alterations in bronchoalveolar lavage cytokines and growth factors | Baseline, 21 days
  Measured by multiplex ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tighe, MD, Principal Investigator — Duke University
Locations (1):
- Duke Asthma, Allergy, and Airway Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No